CLINICAL TRIAL: NCT03091088
Title: Efecto de Dos Tipos de Ejercicio físico Para Prevenir la Osteoporosis en Mujeres Postmenopausicas, un Ensayo Clinico Aleatorizado
Brief Title: Effects of Physical Exercise to Prevent Osteoporosis in Postmenopausal Women
Acronym: Osteo_women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, CARMEN GARCÍA GOMARIZ, PhD, PT, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID_OW
Record Dates: First submitted 2017-03-14; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis, Osteopenia; Physical Activity
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): walking at an intense pace
  Interventions: Other: walking at an intense pace
- Experimental (Experimental): osteoporosis specific-oriented training
  Interventions: Other: osteoporosis specific-oriented training

INTERVENTIONS:
Other: walking at an intense pace — Participants walk 6 kilometers in 1 hour at least 3 times per week
  Arms: Control
Other: osteoporosis specific-oriented training — 1 hour of physical activity, 2 times per week, based on the Asociación Española con la Osteoporosis y la Artrosis (AECOS) recommendations. Sessions are divided in 15 minutes of warmup (8 to 10, 60-second exercises), 30-35 minutes of combined exercises with loads and weights, as well as high intensity exercises, and 10-15 minutes of cooldown activities (based on Frederick relaxation techniques)
  Arms: Experimental

SUMMARY:
According to the World Health Organization criteria, osteoporosis was defined as a bone mineral density that lies 2.5 standard deviations or more below the average value for young healthy women. Osteoporosis is a major cause of fractures and can lead to serious complications in postmenopausal women. For this reason, approaches to prevent the appearance and progression of osteoporosis are of primary importance. This randomized clinical trial analyzes the effects of two types of physical exercise oriented to prevent osteoporosis in postmenopausal women with pharmacological supplements of Calcium and Vitamin-D.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* Pharmacological treatment (VitaminD+Calcium)

Exclusion Criteria:

* Disease or physical-mental condition which prevents to perform the proposed physical exercise

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Femoral neck T-score | Change from baseline score at two years
  The score compares femoral neck bone mineral density to a reference mean
Lumbar spine T-score | Change from baseline score at two years
  The score compares lumbar spine bone mineral density to a reference mean

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Gomariz C, Blasco JM, Macian-Romero C, Guillem-Hernandez E, Igual-Camacho C. Effect of 2 years of endurance and high-impact training on preventing osteoporosis in postmenopausal women: randomized clinical trial. Menopause. 2018 Mar;25(3):301-306. doi: 10.1097/GME.0000000000001005. PMID 29040219